CLINICAL TRIAL: NCT01445002
Title: Safety and Dose Finding Study Based on the Effects of Three Subcutaneous Injections of BM32, a Recombinant Hypoallergenic Grass Pollen Vaccine, on Responses to Allergen Challenge by Skin Testing and in the Vienna Challenge Chamber (VCC) as Well as Immunological Response in Subjects Know to Suffer From Grass-pollen Induced Allergic Rhinitis
Brief Title: Safety and Dose Finding Trial of BM32 in Subjects Suffering From Grass Pollen Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomay AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS-BM32-002; 2011-003368-64 (EudraCT Number)
Record Dates: First submitted 2011-09-26; First posted 2011-10-03 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Grass Pollen Allergy
Keywords: grass pollen allergy; immunotherapy; recombinant vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BM32 low dose (Experimental): 3 subcutaneous injections of 10 micrograms in a time span of 8 weeks
  Interventions: Biological: BM32
- BM32 medium dose (Experimental): 3 subcutaneous injections of 20 micrograms in a time span of 8 weeks
  Interventions: Biological: BM32
- BM32 high dose (Experimental): 3 subcutaneous injections of BM32 over a time span of 8 weeks
  Interventions: Biological: BM32
- Placebo (Placebo Comparator): 3 subcutaneous injections over a time span of 8 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BM32 — Subcutaneous injection of 10 micrograms each of the BM32 components adsorbed on 0.3 mg of aluminum hydroxide every 4 week for a total of 3 injections
  Arms: BM32 low dose
Biological: BM32 — Subcutaneous injection of 20 micrograms of each of the BM32 components adsorbed on 0.6 mg of aluminum hydroxide every 4 weeks for a total of 3 injections
  Arms: BM32 medium dose
Biological: BM32 — Subcutaneous injection of 40 micrograms of each of the BM32 components adsorbed on 1.2 mg of aluminum hydroxide every 4 weeks until a total of 3 injections
  Arms: BM32 high dose
Biological: Placebo — Subcutaneous injection of 1.2 mg of aluminum hydroxide suspension every 4 weeks until 3 injections
  Arms: Placebo

SUMMARY:
The study will evaluate the dose response of immunotherapy against grass pollen allergy using the recombinant grass pollen vaccine BM32. Efficacy will be analyzed by:

* skin prick testing
* grass pollen inhalation challenge
* antibody responses. In addition, the safety of subcutaneous application of BM32 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* History of seasonal allergic rhinitis from grass pollen
* Normal electrocardiogram
* Moderate to severe response to approx. 1500 grass pollen grains/m3 after 2 hrs of exposure in challenge chamber
* Positive skin prick test for grass pollen at or within 12 months preceding screening visit
* Positive RAST (class 2 or higher) for timothy grass pollen and to rPhl p 1 + rPhl p 5 at or within 12 months preceding screening visit

Exclusion Criteria:

* Pregnant or lactating females
* Females with childbearing potential not using medically acceptable birth control
* Structural nasal abnormalities, nasal polyposis, history of frequent nosebleeds, recent nasal surgery or ongoing upper respiratory tract infection
* Any respiratory disease other than mild asthma controlled with occasional short acting beta agonists and normal lung function
* Current or recent participation in another clinical trial
* SIT for grass pollen allergy in the last two years prior to study
* Past or present disease, which may affect outcome of the trial, judged by investigator
* Autoimmune diseases, immune defects including immunosuppression, immune- complex immunopathies
* Suspected hypersensitivity to any ingredients of study medication
* Use of prohibited medication prior to screening and throughout study
* depot corticosteroids (12 weeks)
* oral corticosteroids (8 weeks)
* inhaled corticosteroids (4 weeks)
* Allergic symptoms at the time of screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Minimum effective dose for reduction of total nasal symptom score (TNSS) after inhalation challenge with grass pollen | Baseline and 14 weeks
  Difference in the total Nasal Symptom Score (TNSS) between spending 6 hrs in the Vienna Challenge Chamber (VCC) at screening and spending 6 hrs in the VCC four weeks after the last subcutaneous injection of BM32.

SECONDARY OUTCOMES:
Minimum Effective dose for reduction of Total Non-Nasal Symptom Score (TNNSS) following inhalation challenge with grass pollen | Baseline and 14 weeks
Minimum effective dose for reduction of Global symptom Score upon inhalation challenge with grass pollen | Baseline and 4 weeks after final s.c. injection
Minimum effective dose for reduction of nasal airflow resistance after inhalation challenge with grass pollen | Baseline and 14 weeks
Minimum effective dose to reduce skin reaction to grass pollen allergen upon skin prick testing | Baseline and 14 weeks
Difference in FEV1 and FEV/FVC between screening and completion of vaccination | Baseline and 14 weeks
Frequency of local reactions to treatment | average of 8 weeks from 1st to last injection
Change in allergy specific total IgG | Baseline and average of 12 weeks after randomization
Change in allergy specific IgE | Baseline and average of 12 weeks after randomization
Frequency of systemic reactions to treatment | average of 8 weeks from 1st to last injection
Severity of local reactions to treatment | Average of 8 weeks from 1st to last injection
Severity of systemic reactions to treatment | Average of 8 weeks from 1st to last injection
Frequency of adverse events | average of 14 weeks from 1st injection

CONTACTS AND LOCATIONS:
Locations (1):
- Allergy Center Vienna West, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Zieglmayer P, Focke-Tejkl M, Schmutz R, Lemell P, Zieglmayer R, Weber M, Kiss R, Blatt K, Valent P, Stolz F, Huber H, Neubauer A, Knoll A, Horak F, Henning R, Valenta R. Mechanisms, safety and efficacy of a B cell epitope-based vaccine for immunotherapy of grass pollen allergy. EBioMedicine. 2016 Sep;11:43-57. doi: 10.1016/j.ebiom.2016.08.022. Epub 2016 Aug 20. PMID 27650868